CLINICAL TRIAL: NCT04371497
Title: Three-year Retrospective Study on the Switch From Rapid-acting Insulin Analog to Concentrated U-500 Regular Insulin in Insulin-resistant Type 2 Diabetes Patients Treated by Pump Therapy
Brief Title: Switch From U-100 Insulin Analog to U-500 Regular Insulin in Pumps for Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CHU 20-504
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Insulin Resistance; Continuous Subcutaneous Insulin Infusion; Insulin Pump; Concentrated Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to perform a 3-year retrospective analysis from a cohort of patients with type 2 diabetes that were treated by a pump device and were uncontrolled despite high U-100 insulin requirements. The study reports outcomes after the switch from U-100 U/ml Rapid-Acting Analog to U-500 U/ml Regular Insulin, both administered by Continuous Subcutaneous Infusion.

DETAILED DESCRIPTION:
This study is a retrospective evaluation of a cohort of patients with Type 2 Diabetes from six French centers, who were previously treated by insulin pump therapy, and then switched from U-100 Rapid Acting Insulin analog to 500 U/mL Regular Insulin (Eli Lilly Inc, France) between June 2011 and September 2017. All participants had been previously treated by Multiple Daily Insulin injections and then had been treated by Continuous Subcutaneous Insulin Infusion with U-100 Rapid Acting Insulin analog administered by an insulin pump. Patient's selection criteria included an insulin-resistant state defined by a Total Daily insulin Dose greater than 100 U per day, and a switch from U-100 Rapid Acting Insulin analog to 500 U/mL Regular Insulin during the study period. Data collection from patient medical records included HbA1c, lipid levels, weight, Total Daily insulin Dose, and the recordings of hypoglycemia episodes. Outcomes were recorded at different timelines including baseline and 6, 12, 24 and 36-months after the switch from U-100 to U-500 insulin. Blinded continuous glucose monitoring (CGM) (ipro2, Medtronic Inc., USA) was analyzed in a subgroup of patients having CGM data available at baseline on U-100 insulin and after 6-months on U-500 insulin.

ELIGIBILITY:
Inclusion Criteria:

* T2D diabetes
* Pump therapy with U-100 U/ml rapid-acting analog prior to initiation of U-500 U/ml insulin
* Total daily Insulin dose > 100 U per day

Exclusion Criteria:

* follow up < 3 months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes, treated by pump therapy with U-100 U/ml rapid-acting analog, with a Total daily Insulin dose > 100 U per day, willing to switch to U-500 U/ml insulin administered by Pump
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
differential HbA1c before and after insulin switch | baseline, 1-year, 2-years, 3-years
  HbA1c comparison between baseline and 1, 2, 3 year(s) after the switch to U-HbA1c comparison between baseline and 1, 2, 3 year(s) after the switch to U-500 insulin

SECONDARY OUTCOMES:
Total Daily Insulin Dose | baseline, 1-year, 2-years, 3-years
  Total Daily Insulin Dose at baseline and 1, 2, 3 year(s) after the switch to U-500 insulin
Body Weight | baseline, 1-year, 2-years, 3-years
  Body Weight measured at baseline and 1, 2, 3 year(s) after the switch to U-500
Lipids | baseline, 1-year, 2-years, 3-years
  Plasma Lipids measured at baseline and 1, 2, 3 year(s) after the switch to U-500
Hypoglycemia events | baseline, 1-year, 2-years, 3-years
  Episodes of Hypoglycemia recorded before and during the study
Continuous Glucose Monitoring before and after insulin switch | baseline, 6-month
  Continuous Glucose Monitoring comparison between baseline and 6-month after the switch to U-500

IPD SHARING:
Plan to Share IPD: No